CLINICAL TRIAL: NCT03634111
Title: The Transversus Abdominis Plane Block
Brief Title: The Effect of the Transversus Abdominis Plane Block to Postoperative Analgesia for Cesarean Section
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11-2017/CN-HĐĐĐ
Record Dates: First submitted 2018-08-12; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Obstetric Pain
Keywords: transversus abdominis plane block (TAP block); postoperative analgesia; cesarean section
MeSH Terms: conditions — Labor Pain | interventions — Morphine; Analgesics, Opioid; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Transversus abdominis plane block under the ultrasound guidance
Masking Description: Participants were cesarean section with general anesthesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T group (Active Comparator): The TAP block group was called T group. The participants were performed TAP block under guidance at the end of surgery.
  Interventions: Procedure: TAP block; Drug: Morphine; Drug: Ropivacaine
- C group (Placebo Comparator): The controlled group was called C group. The participants has not TAP block and were treated postoperative analgesia with intravenous morphine to patients controlled analgesia
  Interventions: Drug: Morphine; Drug: Ropivacaine

INTERVENTIONS:
Procedure: TAP block — TAP block was performed under guidance with 0.25% ropivacaine 20 ml each side.
  Other Names: Transversus abdominis plane block
  Arms: T group
Drug: Morphine — Single dose was 1 mg. The locked time was 6 minutes. The limited dose was 40 mg/ 4 giờ.
  Other Names: Opioids
Drug: Ropivacaine — Ropivacaine 0.25% 20 ml each side
  Other Names: Anaropin

SUMMARY:
The transversus abdominis plane block (TAP block) has effect to postoperative analgesia for cesarean section with spinal anesthesia but it was limited for cesarean section with general anesthesia. The hypothesis that this technique has effect to postoperative analgesia for cesarean section with general anesthesia and it could reduce 50% of total morphine consumption during 24 hours after surgery.

DETAILED DESCRIPTION:
This is a randomized, controlled, no-blind clinical trial. The investigators selected 60 cases, who were cesarean section under general anesthesia, age from18 years, and American Society Anesthesiologists (ASA) classification was from II-III. The cases of acute fetal impairment, local anesthesia contraindication, tolerance opioids, liver failure, renal failure, and spinal anesthesia failure were excluded. All cases were randomized assigned two groups: the TAP block group (T group) and controlled group (C group). Each group has 30 cases. The TAP block was performed under the ultrasound guidance with 0.25% of ropivacaine 20 ml each side. The both groups was treated postoperative analgesia with intravenous morphine to patients controlled analgesia (PCA). The primary outcome was total morphine consumption during 24 hours after surgery. The secondary outcomes were the time of required the first dose of morphine, pain score, the complications of TAP block, the side effects of morphine, and satisfaction score of participants. Data was described and analyzed with SPSS 25.0. The sample size was calculated with the hypothesis that TAP block could reduce 50% of dose morphine during 24 hours after surgery, 80% of power, 10% of loss, and 0.05 of alpha error.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section with general anesthesia.
* The ASA classification was from II to III

Exclusion Criteria:

* The acute fetal impairment.
* The severe live or renal failure.
* Tolerance opioids

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption during 24 hours | 24 hours
  Morphine was intravenous perfusion to participants during 24 hours with patients controlled analgesia (PCA).

SECONDARY OUTCOMES:
The time required the first of dose of morphine (hours) | 24 hours
  The time was from the end of surgery to the participants required the first of dose of morphine with PCA.
Pain score: VAS | 24 hours
  Pain score was measured with visual analogue scale (VAS). VAS is from 0 to 10. The zero is complete non-pain and the ten is severe pain
The rate of complications of TAP block | 24 hours
  There were rate of systemic toxicity, puncture peritonea, and hematomae in abdominal wall
The rate of side effect of morphine | 24 hours
  There were rate of sedation, respiratory failure, nause and vomiting, pruritus
The satisfaction of participants: Likert | 24 hours
  It was evaluated with Linkert score. Likerk score is from 1 to 5: 1-strongly disagree, 2-disagree, 3-neither agree nor disagree, 4-agree, 5-strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: THANG T Nguyen, Mr, Principal Investigator — Gia Dinh People Hospital
Locations (1):
- THANG Nguyen Trong, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No